CLINICAL TRIAL: NCT05800483
Title: Improving Decision-Making for Low Health Literate Prostate CA Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 15-192
Record Dates: First submitted 2023-03-08; First posted 2023-04-05 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-03

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healium (Experimental): Healium is a web-based platform that employs a user-centric design and aims to appeal to a low health literate population. It features a simple language and layout, a large font size, contrasting text and background colors, bright color palette, and use of short labels and headings to describe content.
  Interventions: Behavioral: Healium
- Comparison (Healing Choices) (No Intervention): The Healing Choices program represents a virtual health center that patients visit to obtain disease and treatment-related information. The software was designed to be open to exploration with an intuitive layout, without restrictions in terms of order of access. Information is stored in virtual rooms, such as a library, a conference room showing videos by survivors who discuss their approach to treatment, and physician offices containing videos of physicians representing different treatment specialties. All information was extensively vetted by health education experts of the National Cancer Institute's Cancer Information Services (CIS).

INTERVENTIONS:
Behavioral: Healium — web-based platform to elicit patients' preferences about prostate cancer treatment and designed for low health literature populations
  Arms: Healium

SUMMARY:
This study used a randomized controlled trial to evaluate whether Healium (designed to target preference elicitation) is as efficacious as Healing Choices (a comprehensive education and decision tool) in improving outcomes for decision-making and emotional quality of life.

DETAILED DESCRIPTION:
Background: Elicitation of patients' preferences is an integral part of shared decision making, the recommended approach for prostate cancer decision making. However, existing decision aids for this population do not specifically focus on patients' preferences. Healium is a brief interactive web-based decision aid that aims to elicit patient's treatment preferences and is designed for a low health literate population. This study used a randomized controlled trial to evaluate whether Healium (designed to target preference elicitation) is as efficacious as Healing Choices (a comprehensive education and decision tool) in improving outcomes for decision-making and emotional quality of life.

Method: Patients diagnosed with localized prostate cancer who had not yet made a treatment decision were randomly assigned to the brief Healium intervention or Healing Choices, an extensive decision aid previously developed by our group that serves as a virtual information center on prostate cancer diagnosis and treatment. Assessments were completed at baseline, 6-weeks and 3-months post-baseline, and included decisional outcomes (decisional conflict, satisfaction with decision, preparation for decision-making), and emotional quality of life (anxiety/tension and depression), along with demographics, comorbidities, and health literacy.

ELIGIBILITY:
Inclusion Criteria:

* a diagnosis of localized prostate cancer and eligible for all treatment options (ie., surgery, radiation, active surveillance);
* had not yet made a treatment decision or begun treatment; and
* have basic proficiency (grade school level) in reading English.

Exclusion Criteria:

• none

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — required to have a prostate, as this research was on prostate cancer
Enrollment: 327 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Decisional Conflict Scale | 6 weeks post-baseline
  Decisional Conflict was measured with the Decisional Conflict Scale (DCS), a well-validated scale consisting of 16 items that assess four dimensions: informed, clarity, uncertainty, and support. The response ranges are on a 5-point Likert scale ranging from strongly agree to strongly disagree. To come up with a total score, the 16 items are summed, divided by 16 and multiplied by 25. Scores range from 0 (no decisional conflict) to 100 (extremely high decisional conflict).
Decisional Conflict Scale | 3 months post-baseline
  Decisional Conflict was measured with the Decisional Conflict Scale (DCS), a well-validated scale consisting of 16 items that assess four dimensions: informed, clarity, uncertainty, and support. The response ranges are on a 5-point Likert scale ranging from strongly agree to strongly disagree. To come up with a total score, the 16 items are summed, divided by 16 and multiplied by 25. Scores range from 0 (no decisional conflict) to 100 (extremely high decisional conflict).

SECONDARY OUTCOMES:
Profile of Mood States- Short form | 6 weeks post-baseline
  The Profile of Mood States (POMS) is a psychological rating scale used to assess transient, distinct mood states. It is made of subscales for depression, tension, fatigue, confusion, anger, vigor and esteem-related affect. It consists of 30 items, each measured on a 5-point scale ranging from "not at all" to "extremely". A total score is calculated by summing the totals for the negative scales and subtracting the totals for the positive scales.
Profile of Mood States-Short form | 3 months post-baseline
  The Profile of Mood States (POMS) is a psychological rating scale used to assess transient, distinct mood states. It is made of subscales for depression, tension, fatigue, confusion, anger, vigor and esteem-related affect. It consists of 30 items, each measured on a 5-point scale ranging from "not at all" to "extremely". A total score is calculated by summing the totals for the negative scales and subtracting the totals for the positive scales.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Northwell Health, Manhasset, New York
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Diefenbach MA, Marziliano A, Tagai EK, Pfister H, Lapitan E, Hall SJ, Vira M, Ibrahim S, Aibel K, Kutikov A, Horwitz EM, Miyamoto C, Reese AC, Miller SM. Preference Elicitation and Treatment Decision-Making Among Men Diagnosed With Prostate Cancer: Randomized Controlled Trial Results of Healium. J Med Internet Res. 2023 Oct 20;25:e46552. doi: 10.2196/46552. PMID 37862103